CLINICAL TRIAL: NCT04945759
Title: Comparison of the Efficacy of Russian and Aussie (Australian) Currents With Isokinetic Exercise in Individuals With Patellofemoral Pain Syndrome: A Randomized Controlled Study.
Brief Title: Comparison of the Efficacy of Russian,Aussie Currents With Isokinetic Exercise Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, MUSA ÇANKAYA MSc.PT, Master of Science (Lecturer), Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11.02.2020 V;1
Record Dates: First submitted 2021-05-22; First posted 2021-06-30 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Aussie Current
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Posttest and control grouped randomized controlled clinical trial.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Isokinetic Exercise (İE) Group: (Experimental): Isokinetic Exercise (IE) Group:
  (Knee Joint Flexion / Extension, Hip Joint Internal / External Rotation and Abduction / Adduction Strengthening Program)
  Patients will be seated on the isokinetic Cybex-Humac Norm device in a 90° upright sitting position. It will be fixed to the seat with torso, pelvis and thigh straps. During this training, patients will be told that the dynamometer arm will bring the knee from extension to flexion. During this exercise, the patient will be advised to resist the dynamometer as much as possible while moving the knee in flexion/extension, internal/external rotation, and abduction/adduction with the dynamometer.
  Interventions: Device: Isokinetick Exercise, Aussie Current, Russion Current, Plasebo Electirical Stimulasyon
- Isokinetic Exercise + Aussie Current (IE+AC)Group: (Active Comparator): Aussie Current and Isokinetic Exercise program will be applied to the patients. The distal electrode is placed on the anterior part of the thigh and superior to the patella. The proximal electrode will be placed on the thigh. One electrode will be placed between the anterior superior and posterior superior iliac spine of the PFPS(Patellofemoral Pain Syndrome) side and the other electrode will be placed in a triangle on the greater trochanter of the femur in the gluteus medius muscle. By contacting the Turkish authorities of the BTL 4825SPREMIUM device, the current was adjusted in the Aussie Current 1 kHz frequency, 400 ms phase time, 50 hz burst frequency, 4 ms duration device. This new burst modality medium frequency alternating current will be applied to the patient for 20 minutes.
  Interventions: Device: Isokinetick Exercise, Aussie Current, Russion Current, Plasebo Electirical Stimulasyon
- Isokinetic Exercise + Russian Current (IE+RC) Group: (Active Comparator): Isokinetic Exercise program will be applied to the patients. Similarly, as with the Aussie Current, the Russian current will be applied to the vastus lateralis-medialis and gluteus medius muscles.
  Russian current will be set as 2500 Hz sinusoidal current, 200 ms phase time, 50 hz burst frequency, 50% duty cycle, 10 ms duration.
  The patient will be treated for 20 minutes.
  Interventions: Device: Isokinetick Exercise, Aussie Current, Russion Current, Plasebo Electirical Stimulasyon
- Isokinetic Exercise + placebo Electrical Stimulation (IE+PES) Group: (Placebo Comparator): Isokinetic Exercise program will be applied to the patients. The appropriate modalities will be set on the electrical stimulation device, but the device will not operate. It will be applied for 20 minutes.
  Interventions: Device: Isokinetick Exercise, Aussie Current, Russion Current, Plasebo Electirical Stimulasyon

INTERVENTIONS:
Device: Isokinetick Exercise, Aussie Current, Russion Current, Plasebo Electirical Stimulasyon — Evaluation and treatment will be done with the Cybex humac device.

SUMMARY:
Summary

Patellofemoral pain syndrome (PFPS) is defined as common anterior knee pain that occurs during non-traumatic activities such as squatting, running, climbing and climbing stairs.The effectiveness of electrotherapy in increasing muscle strength and endurance in PFPS has generally been investigated using low frequency electrical stimulation methods, and studies on the effectiveness of medium frequency burst module alternating currents are few in number. Since there are no studies in the literature comparing the efficacy of Russian and Aussie currents from mid-frequency burst modulated alternating currents with isokinetic exercise in patients with PFPS, the aim of this study is to examine the pain, functionality, daily living activities of Russian and Aussie currents with knee and hip Isokinetic Exercise (IE) in patients with PFPS and its effect on quality of life.

This study, which has a randomized controlled and single-blind design, is planned to be conducted on at least 60 volunteers who meet the inclusion criteria of patients with PFPS who came to Necmettin Erbakan University Sports Medicine Clinic. Participants' physical and socio-demographic information will be recorded; pain intensity Patellofemoral Syndrome Pain Severity Scale; functionality Kujala Patellofemoral Score, Timed Up and Go Test and stair climb test; activity levels Tegner Activity Level score; functional impairment Lysholm Knee Scoring Scale; activities of daily living Knee Test for Activities of Daily Living; quality of life Short Form SF-36; passive and painless active range of motion goniometer; Isokinetic forces of quadriceps, hamstring and gluteus medius muscles CYBEX (2009) device; The Q angle will be evaluated using a goniometer.

Participants will be randomized into four groups; The first group will receive knee and hip IE treatment for three weeks for 15 sessions, the second group will receive Aussie Current in addition to IE, the third group will receive Russian Current in addition to IE, and the fourth group will receive placebo electrical stimulation in addition to IE. Evaluations will be made at the beginning, immediately after the first treatment, at the end of three weeks of treatment and one month after the end of the treatment, in total four times. It is thought that the results of the study will be an important source of information about the place of medium frequency burst modulated alternating currents in physiotherapy programs of patients with PFPS.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is the most common pain syndrome of the knee arising around the patella due to knee overload during flexion and extension. It is defined as common anterior knee pain that occurs during non-traumatic activities such as squatting, running, climbing and climbing stairs. Risk factors for PFPS include dynamic valgus, female gender, foot abnormalities, overuse and sudden increase in physical activity, patellar instability, and quadriceps weakness .

In order to reveal effective treatment in PFPS, primary reasons that may cause the syndrome should be emphasized. The causes of PFPS are multifactorial and it is difficult to determine the actual effects that may cause the disease.However, when PFPS is considered from a biomechanical point of view, there is a strong relationship between the knee joint and the ankle and hip joint.

While rest, ice and analgesics are used in the early period in PFPS treatment, non-steroidal anti-inflammatory drugs (NSAIDs), patellar banding, patellofemoral knee and foot orthoses, biofeedback, running gait retraining, blood circulation restriction therapy are used in the treatment of PFPS in the early period. Dry needling, manual therapy, biophysical agents, patient education and combined therapies are used. In the treatment of patellofemoral pain syndrome, the treatment method that has been focused in recent years is conservative treatment. Among these, physiotherapy is the cornerstone of treatment.

Although the common treatment is quadriceps strengthening, in recent years, therapies have been emphasized to strengthen the gluteus medius and increase the stability of the core. At the 5th International Meeting of the Patellofemoral Pain Research Center (2018, Australia), combined strengthening programs with strengthening of the quadriceps and hip muscles were recommended in the treatment of PFPS.

Although a versatile treatment is generally performed, the rate of PFAS recurrence is 91%. Due to the high recurrence rate, more effective treatment options should be revealed. When the literature is reviewed, it has been reported that in PFPS cases, there is an increase in muscle strength and endurance with the isokinetic exercise (IE) program, and this provides dynamic knee stabilization.The IE program is mostly in the direction of knee flexion / extension, and it has been found that there are very few applications of IE programs in the direction of hip (gluteus medius) abduction / adduction, internal and external rotation.

Physiotherapy applications are directed towards the management of developing dysfunction and reducing pain. Strengthening and endurance training are emphasized in routine treatment. Although isokinetic enhancement programs are the most effective method in treatment, neuromuscular electrical stimulation rehabilitation programs are also frequently used. The effectiveness of eletrotherapy modalities to increase muscle strength and endurance is not clear. Among these, medium frequency burst modality alternative (Russian and Australian) current can be used as a new treatment option. Low frequency pulsed currents (LFPC) and medium (kHz) frequency alternating currents (FAC) are frequently used in physiotherapy and rehabilitation.

Austrian current (AC) is a more effective and comfortable current between 1-10 kHz medium frequency currents. This current can be used for various purposes including muscle strengthening, pain control, increasing circulation, edema control and aesthetic treatments.

AC started to be used in the Latin America region with the devices it launched with Ibramed company in 2010. It creates much less discomfort in the patient compared to AC Russ Current (RC) and low frequency currents. It is used in sinusoidal wave form.

In recent meta-analysis studies on PFAS, she stated that new methods should be aimed at identifying the most cost-effective and most effective treatment modalities. Although there are studies in the literature showing the effect of neuromuscular electrical stimulation, it has been found that there are no studies comparing medium frequency burst modulated alternating currents (AC and RC) with IE in patients with PFPS.

In the national literature, there are no scientific studies on the Australian current method. The application of RC and AC together with the isokinetic method, whose effectiveness has been determined in the literature, is very important in terms of determining the most effective treatment method.

Objectives of the study In individuals with PFPS, isokinetic IE together with medium frequency burst modality alternating currents;

* To reduce the pain during rest and activity,
* Increasing functional mobility,
* Facilitating Activities of Daily Living (FADL),
* To increase the quality of life.

Sample of the Research Power analysis G*Power 3.1.9.2 program was used to calculate the sample size. The power of the research is defined as the possibility of revealing the difference between the two applications. The effect size was 0.25, the alpha level was 0.05, and the power of the study was 0.95, and it was determined that a total of 52 subjects should be included in the study in the calculation made in the form of four groups and four repeated measurements made in the G-power program. In similar studies in the literature, it was determined that there was a 15% loss. In this study, it was planned that a total of 60 cases should be included in the study, assuming 15% loss.

Application Closed opaque envelopes showing the patient's group will be prepared. Opaque envelopes will be listed from 1 to 60 according to the randomly generated numbers. An envelope will be given to the patient according to the order of the incoming patient. The assignment code of each patient will only be disclosed to the physiotherapist performing the treatment at the beginning of the treatment protocol.The physiotherapist will include the patient in the group in accordance with the code and perform the application.It will be ensured that subjects in the RC, AC and placebo electrical stimulation groups do not know what type of stimulation they were given.

Pilot Study A pilot study will be conducted on a group of four people (one person from each group) in order to evaluate the applicability of data collection forms and treatments to be used in the study.

Blinding İsokinetic exercise (IE), Aussie current (AC), Rus current (RC), Placebo Electrical Stimulation (PES) Group,

Patients in theIE, IE + AC, IE + RC, IE +PEC groups will not be informed about the application other than exercise. The evaluations will be carried out by a physiotherapist who does not know which group the patients are in.

The physical (age, height, gender, body mass index) and socio-demographic (occupation, marital status, educational status, income-expense balance) information of the participants who will read the informed consent form and volunteer to participate in the study will be recorded. The duration of the PFPS complaint (weeks), the time elapsed since the diagnosis of PFPS (weeks), history characteristics (hypertension, diabetes mellitus and other chronic systemic diseases) will be noted. Pain intensity at rest and during performance-based functional mobility tests will be determined using the Patellofemoral Syndrome Pain Severity Scale (PSPSS). All evaluations will be done before treatment (BT), immediately after treatment, after three weeks of treatment (TA), and one month after treatment (Control).

Treatment Program The Isokinetic Exercise program will be applied to the patients as described above. Appropriate modalities will be set on the electrical stimulation device, but the device will not be operated. It will be applied for 20 minutes.

4 treatment groups will be treated five days a week, 15 sessions for three weeks. If participants miss any treatment, there will be additional treatment sessions.

Dependent Variables of the Research

* Patellofemoral Syndrome Pain Severity Scale
* Timed Get Up and Go Test result
* Stair up and down test
* Kujala Patellofemoral score
* Tegner Activity Level score
* Lysholm Knee Scoring Scale score
* Knee Test Score for Daily Living Activities
* Short Form SF-36 score
* Passive and Painless Active Knee Joint Range of Motion
* Isokinetic Muscle Strength score
* Q Angle Measurement Degree

Study Independent Variable

* Isokinetic Exercise Therapy Program
* Isokinetic Exercise Australia Current Therapy Program
* Isokinetic Exercise Russian Current Therapy Program
* Isokinetic Exercise Placebo Electrical Stimulation Therapy Program

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-55,
* Being able to read and write in Turkish,
* Having pain for more than a month,
* Having anterior knee pain without trauma,
* To have a pain intensity of three points and / or above according to the Visual Analogue Scale (VAS) in the peri or retropatellar region in the previous week.

Exclusion Criteria:

* Meniscus, cross and collateral ligament, iliotibial band lesion, Having pes anserin tendinitis, Osgood-Schlatter syndrome,
* Sinding-Larsen-Johansson Syndrome, previous patellar dislocation and previous knee surgery, having received knee injection treatment at least three months ago,
* Using Nonsteroidal Anti-inflammatory and Cortisone drugs frequently once a week or more,
* Trauma history and neurological disease,
* Having a patellar fracture, osteoarthritis or other intra-articular knee pathology,
* Having pain and knee effusion reflected from the hip and lumbar region (
* Those with contraindicated conditions for electrical stimulation (biomedical device implant, pregnant women, neuropathy, muscle abnormalities or hypersensitivity, malignancy, hemorrhagic area, skin damage, active infection in the area where the electrodes are placed) (3,59).

Having had previous electrical stimulation therapy

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Patellofemoral Syndrome Pain Severity Scale | 3 minute
  It is a scale consisting of 10 parameters that evaluates the pain in the activities of the individual during the last week with VAS. These activities include climbing stairs, crouching on the ground, walking, jogging, fast jogging, participation in a sport, sitting with bent knees, kneeling, resting and sleeping, resting after activity. Individuals will also mark activities they did not do in the last week as "I did not do". The maximum score is 100 and the evaluation results will be recorded in%.
Kujala Patellofemoral Score | 3 minute
  The Turkish validity and reliability study was conducted by Kuru et al. KPS includes questions about patellar alignment and the position of the patella, and consists of 13 items that evaluate subjective responses to specific activities and symptoms thought to be associated with PFAS. It is scored from a minimum of 0 to a maximum of 100 points. A variation of 8-10 points constitutes the minimum significant difference in clinical practice. Lower scores indicate more pain and disability, while higher scores indicate fewer disabilities. In the guideline published by the American Physical Therapy Association, Orthopedic Physical Therapy Academy, it was stated that the use of KPS form in PFAS patients reveals high quality data.
Knee Test for Daily Living | 3 minute
  Symptoms and functional limitations of individuals in daily living activities will be evaluated with the Knee Test for Daily Living Activities (KOS-ADLS), which is a valid and reliable questionnaire that has been made in Turkish. The test includes six questions about symptoms: pain, stiffness, swelling, relaxation / flexion of the knee, weakness, and limping. It also includes eight questions about functional limitations, including walking, climbing stairs, descending stairs, standing, kneeling, crouching, sitting with bent knees, and getting up from a chair. The test is scored between 0-5. The patient's scores from each question are added up and the total score is divided by 70 and multiplied by 100.
A)Measurement of Isokinetic Muscle Strength of Knee Flexion / Extension: | 8 minute
  Measurement of Isokinetic Muscle Strength:
  Before the test, patients will be warmed up for 10 minutes with an elliptical bicycle (the brand of the device). Isokinetic muscle strength of the quadriceps and Hamstring groups (at 60°/120°/180 °/second velocity) will be measured using Humac Norm System.
  To familiarize patients unfamiliar with the test, 3 sub-maximal contractions and 1 maximal contraction will be performed for each muscle group and at each speed. The affected extremity will be evaluated for testing. After the test, the flexor and extensor peak torques at 60°/120°/180° second angular velocities and the work done and hamstring/quadriceps (H/Q) ratios will be calculated in the computer environment. Peak torque values will be recorded.
Interna /External Rotation Measurement of Isokinetic Hip Strength: | 5 minute
  In addition, taking into account the points in the evaluation of hip flexion/extension using the Cybex Humac Norm System, the patient will be positioned in the sitting position with the knee and hip at 90° flexion, and the trunk at 30° extension.
  The hip on the tested side will be fixed over the thigh, and the leg area will be fixed with a band just above the ankle. The dynamometer axis will be aligned with the long axis of the patella. The test will begin from maximum active external rotation to internal rotation. Hip medial and lateral rotation will be applied at speeds of 30°/60° seconds. 30 seconds of rest will be given after each speed. The test will be performed after four submaximal repetitions at each rate. Peak torque, internal/external force, internal/external torque ratio will be calculated.
Abduction/Adduction Measurement of Isokinetic Hip Strength: | 2 minute
  The cases will be placed on the Cybex Humac Norm System. The non-tested knee and hip (table side) will be fixed with a tape.
  The pelvis will be fixed on the CYBEX system with a pelvic band. The axis of the extremity to be tested will be aligned 2 centimeters medial and below the anterior superior iliac crest. The lever arm of the dynamometer will be fastened just above the knee with the help of a belt. Gravity correction will be provided with extreme weight during the test. The test will be started in the full abduction position. In addition, hip abduction/adduction will be evaluated at 30°/60° second rates. Four submaximal repetitions at each speed and a fifth test will be performed. Peak torque, abduction/adduction force, abduction/adduction torque ratio will be calculated.

SECONDARY OUTCOMES:
Timed Get Up and Go Test | 2 minute
  It is a test to evaluate dynamic balance and functional mobility. In various populations from children to the elderly; It is used in many conditions including osteoarthritis, joint arthroplasty, rheumatoid arthritis, hip fractures, stroke, vertigo, cerebral palsy. The test will be started with the patient's feet flat on the floor and arms in a standing position on the armrest of the chair. The person is asked to stand up from the chair he is sitting in, walk 3 meters safely and at a normal pace, turn around, walk back, and sit on the chair again. The time is recorded in seconds.
Lysholm Knee Scoring Scale | 2 minute
  It consists of eight subtitles scored differently (limping and used support 5 points, locking 15 points, instability and pain 25 points, swelling 10 points, climbing stairs 10 points and squatting are scored on 5 points. Higher values mean better results: 95-100 points out of 100 points are evaluated as excellent, 84-94 points good, 65-83 points medium and <65 points bad. Cultural adaptation of Lysholm knee score to Turkish Çelik et al. made by, it is stated that it is reliable and valid.
Q Angle Measurement: | 3 minute
  It is the narrow angle formed by a line drawn from the Spina Iliaca Anterior Superior (SIAS) to the midpoint of the patella and the lines drawn from the midpoint of the patella to the midpoint of the tuberositas tibia.
  Goniometers are frequently used in Q angle measurements because of their practicality and low cost. Goniometric Measurement: In this measurement technique, the center of the goniometer is placed in the center of the patella, the fixed arm shows the tibial tubercle and the movable arm shows the SIAS. The measurement can be taken while the person is standing or lying on their back. In standing measurements, the knees should be in extension and equal weight should be applied to both lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: MUSA ÇANKAYA, Msc, Principal Investigator — Necmettin Erbakan University; İLKİM ÇITAK KARAKAYA, Professor, Study Director — Muğla Sıtkı Koçman University; PELİN MELDA YARGIÇ, PhD, Study Director — Necmettin Erbakan University
Locations (1):
- Musa Çankaya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
randomized controlled trial
Supporting Information: Study Protocol
Time Frame: It will be published in a peer-reviewed journal within 6 months after the study is completed.
Access Criteria: The protocol of the research will be published in an international congress as soon as possible. Broadcast link will be shared.